CLINICAL TRIAL: NCT07029854
Title: Laser Acupoints Stimulation on Xerostomia Related Chemoradiotherapy for Head and Neck Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nehal Gamal Ebrahim Elwerish, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005539
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Xerostomia Following Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LASER acupoints therapy + Medical treatment (Experimental): This group will include twenty-seven patients suffering xerostomia (dryness of mouth), who will receive LASER acupoints therapy (3 times per week, for 4 weeks), plus medical treatment.
  Interventions: Other: Medical treatment; Other: LASER acupoints therapy
- Pseudo-LASER acupoints therapy + Medical treatment (Placebo Comparator): This group will include twenty-seven patients suffering xerostomia (dryness of mouth), who will receive pseudo-LASER acupoints therapy plus medical treatment (for 4 weeks).
  Interventions: Other: Medical treatment; Other: Pseudo-LASER acupoints therapy

INTERVENTIONS:
Other: Medical treatment — They will receive oral chemotherapy, based on the cancer stage, and will also undergo radiotherapy.
Other: LASER acupoints therapy — LASER acupoints therapy will use the Pointer Pulse device (GMT2000 s.r.l., Italy), emitting 650 nm red light with an audio trimmer for acupoint detection. Treatment parameters include 5 mW power, 120 s irradiation per point over a 3.14 mm² area (fluence: 19.2 J/cm², power density: 0.16 W/cm², total dose: 0.6 J). Continuous red laser will be applied for effective stimulation. Sessions will occur once weekly for five weeks. Bilateral stimulation will follow this order: left hand, left face, trunk, right face, and right hand. Targeted acupoints: LI 2 Erjian, ST 5 Daying, ST 6 Jiache, ST 7 Xiaguan, SI 19 Tinggong, and BL 13 Feishu.
  Arms: LASER acupoints therapy + Medical treatment
Other: Pseudo-LASER acupoints therapy — For the pseudo-LASER acupoints therapy, the same procedures and sequence of acupoint application will be followed as in the active treatment. However, the Pointer Pulse device (GMT2000 s.r.l., Italy) will be deactivated to emit no therapeutic laser light while maintaining visual and audio cues to mimic real stimulation. The device will appear active to ensure blinding. Sessions will be conducted once weekly for five weeks, applying the probe to the same bilateral acupoints in the following order: left hand, left face, trunk, right face, and right hand. The targeted points will be LI 2 Erjian, ST 5 Daying, ST 6 Jiache, ST 7 Xiaguan, SI 19 Tinggong, and BL 13 Feishu.
  Arms: Pseudo-LASER acupoints therapy + Medical treatment

SUMMARY:
The purpose of the study is to evaluate to effect of LASER acupoints stimulations on xerostomia patients during chemoradiation therapy after head and neck cancer.

DETAILED DESCRIPTION:
The current diagnosis is based on the primary complaint reported by the patient. A previous study found that patients with cancer reported different degrees of dry mouth, reduced drinking and eating and waking up at night due to dry mouth and that the risk of progression to oral ulcers was higher among this patient population and could significantly affect the quality of life.

Acupuncture may be effective in treating xerostomia and also, acupuncture has been shown to increase salivary flow in healthy volunteers.

As xerostomia gradually comes to the attention of the wider medical community, clinical evidence is slowly starting to amass to help assess which treatments are most effective, but more research is needed. Furthermore, there is a lack in the quantitative knowledge and information in the published studies about benefits of acupuncture on xerostomia during chemo radiation therapy. So, this study is designed to outline the therapeutic efficacy of acupuncture on xerostomia during chemo radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Chemoradiation therapy
* Carcinoma in the head and neck area (NPC)
* Anatomically intact parotid and submandibular glands.
* All patients will be clinically and medically stable when attending the study.

Exclusion Criteria:

* They had a history of xerostomia;
* They had suspected or confirmed physical closure of salivary gland.
* ducts on either side.
* They had known bleeding disorders.
* They Were taking heparin or warfarin.
* They had contraindications for the use of acupuncture at any acupoints.
* They had history of cerebrovascular accident or spinal cord injury.
* They had taken any drug or herbal medicine in the past 30 days that could affect salivary function.
* They were planning to, or ended up taking such a substance during the study.
* Any therapy that may affect treatment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-18 (Estimated); Primary Completion 2025-08-18 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Xerostomia Inventory score | 4 weeks
  Participants will complete the Xerostomia Inventory (XI) questionnaire, a validated tool measuring the subjective burden of dry mouth. It consists of 11 items covering symptoms such as dryness of the mouth, lips, eyes, nose, and face, difficulty with dry foods, sipping liquids, sucking sweets, and nighttime thirst. Responses are rated on a 5-point Likert scale from Never (1) to Very Often (5). Total scores are converted to a 0-10 scale, where 0 represents no burden and 10 indicates an excruciating burden. The questionnaire will be administered at baseline and post-treatment.

SECONDARY OUTCOMES:
Stimulated salivary flow rate (SSFR) by Sialometry | 4 weeks
  Sialometry tests will be used to assess salivary flow. Normal stimulated flow ranges from 1.5-2.0 mL/min, and unstimulated flow from 0.3-0.4 mL/min. Hyposalivation will be diagnosed if stimulated flow is below 0.5-0.7 mL/min or unstimulated flow is under 0.1 mL/min. For unstimulated sialometry, patients will be instructed to expel saliva passively into a glass every minute for 6 minutes without swallowing. For stimulated sialometry, patients will consume something sweet and collect saliva every minute for 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Mohamed Abd El Baky, PhD, Study Chair — Professor, Cairo university; Adel Mahmoud Attia, PhD, Study Director — Lecturer, Zagazig university; Doaa Atef Aly, PhD, Study Director — Lecturer, Cairo university
Locations (1):
- El Hussein university Hospital, Cairo, Egypt